CLINICAL TRIAL: NCT03943212
Title: The Effect of Blood Flow Rate on Dialysis Recovery Time in Patients Undergoing Maintenance Hemodialysis - A Prospective, Parallel-Group, Randomized Controlled Trial
Brief Title: The Effect of Blood Flow Rate on Dialysis Recovery Time in Patients Undergoing Maintenance Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Satellite Healthcare (Other)
Responsible Party: Principal Investigator, Brigitte Schiller-Moran, MD, Chief Medical Officer, Satellite Healthcare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR064RT
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: ESRD; Fatigue; Hemodialysis-Induced Symptom
Keywords: Patient-Reported Outcomes; Post-dialysis Fatigue; Dialysis Recovery Time
MeSH Terms: conditions — Kidney Failure, Chronic; Fatigue

STUDY DESIGN:
Intervention Model Description: Parallel-Group, Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Rate Reduction (Experimental): Participants will have their hemodialysis blood flow rate reduced on their regular schedule.
  Interventions: Other: Blood Flow Rate Reduction
- Control (Sham Comparator): Participants will continue to receive regularly-scheduled hemodialysis without any changes to the prescription.
  Interventions: Other: Control

INTERVENTIONS:
Other: Blood Flow Rate Reduction — Hemodialysis blood flow rate will be reduced by 100 mL/min, or to a minimum of 300 mL/min, whichever is higher. Patients will be surveyed regarding their dialysis recovery time and other symptoms weekly.
  Arms: Blood Flow Rate Reduction
Other: Control — No changes will be made to the dialysis prescription. Patients will be surveyed regarding their dialysis recovery time and other symptoms weekly.
  Arms: Control

SUMMARY:
A majority of patients with end-stage renal disease (ESRD) on in-center hemodialysis (HD) require several hours to recover from fatigue after an HD session. Evidence for practical interventions to improve this recovery time from conventional in-center HD is lacking. This study investigates the effects of reducing HD blood flow rates on patients' self-reported post-dialysis fatigue.

DETAILED DESCRIPTION:
Post-dialysis fatigue reduces patients' quality of life and is also associated with cardiovascular events and mortality. Dialysis recovery time (DRT) is a measure of post-dialysis fatigue. Internationally, it has been found that more than a quarter of maintenance HD patients report >6 hours of DRT. The interventions showing the most improvement in DRT involve increases in treatment time, suggesting that post-dialysis fatigue may be in part related to the rate of solute clearance. Solute clearance rate is just one part of extending dialysis time, and its effect on DRT in patients undergoing typical-length dialysis sessions is not known. There is scant evidence to guide blood flow rate prescriptions aside from meeting clearance targets. Blood flow rate reductions are easily-implementable interventions that would slow solute clearance rates and may have an effect on post-dialysis fatigue.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of end-stage renal disease undergoing hemodialysis in the San Francisco Bay Area at approved Satellite Healthcare dialysis centers.
* Dialysis recovery time of 6 or more hours.
* Not hospitalized in the 7 days prior to study

Exclusion Criteria:

* Currently or possibly pregnant, currently trying to become pregnant
* Inability to provide informed consent
* Inability to provide responses to survey questions
* Planned move away from the current hemodialysis center within the study period
* Undergoing nocturnal hemodialysis, planned changed to nocturnal or peritoneal dialysis, planned kidney transplant within the study period, or other major planned change in hemodialysis prescription
* Primary nephrologist objection to enrollment

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Dialysis Recovery Time | 4 weeks
  Mean difference in change in Dialysis Recovery Time between the Blood Flow Rate Reduction group and the Control group. Dialysis recovery time is measured by asking the question, "How long did it take you to recover from dialysis?"

SECONDARY OUTCOMES:
London Evaluation of Illness | 4 weeks
  Mean difference in change in survey responses for measures of quality of life as assessed by the London Evaluation of Illness Tool.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Schiller, MD, Principal Investigator — Chief Medical Officer
Locations (18):
- United States (18):
  - Satellite Dialysis Capitola, Capitola, California
  - Satellite Dialysis Daly City, Daly City, California
  - Satellite Dialysis Gilroy, Gilroy, California
  - Satellite Dialysis Menlo Park, Menlo Park, California
  - Satellite Dialysis Milpitas, Milpitas, California
  - Satellite Dialysis Mountain View, Mountain View, California
  - Satellite Dialysis East San Jose, San Jose, California
  - Satellite Dialysis Santa Teresa, San Jose, California
  - Satellite Dialysis Silver Creek, San Jose, California
  - Satellite Dialysis South San Jose, San Jose, California
  - Satellite Dialysis White Road, San Jose, California
  - Satellite Dialysis Bascom, San Jose, California
  - Satellite Dialysis Stevens Creek, San Jose, California
  - Satellite Dialysis West San Leandro, San Leandro, California
  - Satellite Dialysis San Mateo, San Mateo, California
  - Satellite Dialysis South San Francisco, South San Francisco, California
  - Satellite Dialysis Sunnyvale, Sunnyvale, California
  - Satellite Dialysis Watsonville, Watsonville, California

IPD SHARING:
Plan to Share IPD: No